CLINICAL TRIAL: NCT04829305
Title: A Phase 1, Single Center, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR2285 Single Oral Administration in Healthy Caucasian Participants
Brief Title: A Trial of SHR2285 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHR2285-105
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Three different cohorts can enroll healthy Caucasian participants; males and females in each cohort separately.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose of SHR2285 (Experimental): The subjects will receive a single dose of SHR2285 (cohort 1).
  Interventions: Drug: SHR2285
- Medium dose of SHR2285 (Experimental): The subjects will receive a single dose of SHR2285 (cohort 2).
  Interventions: Drug: SHR2285
- High dose of SHR2285 (Experimental): The subjects will receive a single dose of SHR2285 (cohort 3).
  Interventions: Drug: SHR2285

INTERVENTIONS:
Drug: SHR2285 — SHR2285 is a selective inhibition of human FXIa small molecule compound.

SUMMARY:
This is a phase 1 open-label study

DETAILED DESCRIPTION:
This is a phase 1 open-label study. The objective of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of oral administered SHR2285 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the trial procedures and possible adverse events, volunteers to participate in the trial, and provides written informed consent.
* Be able to comply with all the requirements and able to complete the study.
* Male or female aged between 18 years and 55 years (inclusive) at the date of signed consent form.
* No clinically significant abnormalities in medical history, general physical examination, vital signs, and laboratory tests.
* Men and women of childbearing potential (WOCBP) must agree to take effective contraceptive methods and have no plan to have a child from signing the consent form to 16 weeks after IP administration.

Exclusion Criteria:

* Receipt of any other investigational drugs or medical devices within 3 months prior to screening (according to the date of signed consent form).
* History of illicit or prescription drug abuse or addiction within one year of screening, or positive urine drug screen at screening and Day-1. The urine drug screen may be repeated at the discretion of the investigator and the reason for repeat needs to be documented clearly (e.g., suspicion of false positive due to diet).
* Receipt of any other investigational drugs or medical devices within 3 months prior to screening (from the date of signed consent form).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Adverse events | Start of Treatment to end of study (approximately 7 days)
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics-AUC0-last | Start of Treatment to outpatient (approximately 3 days)
  Area under the concentration-time curve from time 0 to last time point after SHR2285 administration
Pharmacokinetics-AUC0-inf | Start of Treatment to outpatient (approximately 3 days)
  Area under the concentration-time curve from time 0 to infinity after SHR2285 administration
Pharmacokinetics-Tmax | Up to 3 days
  Time to Cmax of SHR2285 and its metabolite SHR164471
Pharmacokinetics-Cmax | Up to 3 days
  Maximum observed concentration of SHR2285 and its metabolite SHR164471
Pharmacokinetics-CL/F | Up to 3 days
  Apparent clearance of SHR2285 and its metabolite SHR164471
Pharmacokinetics-Vz/F | Up to 3 days
  Apparent volume of distribution during terminal phase of SHR2285 and its metabolite SHR164471
Pharmacokinetics-t1/2 | Up to 3 days
  Terminal elimination half-life of SHR2285 and its metabolite SHR164471
Coagulation factor XI (FXI) activity | Up to 3 days
  Coagulation factor XI (FXI) activity
Percentage change of coagulation factor XI (FXI) activity thromboplastin time (APTT) and fold change from baseline | Up to 3 days
  Percentage change of coagulation factor XI (FXI) activity
Activated partial thromboplastin time | Up to 3 days
  Activated partial thromboplastin time
Fold change of activated partial thromboplastin time from baseline | Up to 3 days
  Fold change of activated partial thromboplastin time from baseline
Prothrombin time | Up to 3 days
  Prothrombin time
Fold change of prothrombin time from baseline | Up to 3 days
  Fold change of prothrombin time from baseline
International normalized ratio | Up to 3 days
  International normalized ratio
Fold change of international normalized ratio from baseline | Up to 3 days
  Fold change of international normalized ratio from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jasmine Daisy Williams, Principal Investigator — Study Principal Investigator
Locations (1):
- Linear Clinical research, Perth, Western Australia, Australia